CLINICAL TRIAL: NCT00863681
Title: Long-term Extension, Multicentre, Multi-national Study to Evaluate the Safety and Tolerability of Oral BAY63-2521 (1mg,1.5 mg, 2.0 mg, 2.5 mg Tid) in Patients With Symptomatic Pulmonary Arterial Hypertension (PAH)
Brief Title: BAY63-2521:Long-term Extension Study in Patients With Pulmonary Arterial Hypertension
Acronym: PATENT-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12935; 2008-003610-94 (EudraCT Number)
Record Dates: First submitted 2009-03-13; First posted 2009-03-18 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary arterial hypertension; PH; Stimulator
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Riociguat (BAY63-2521)

INTERVENTIONS:
Drug: Riociguat (BAY63-2521) — BAY63-2521: 1mg tid -2.5 mg tid oral until end of study

SUMMARY:
Patients who have completed the 12 weeks treatment of the PATENT-1 trial (study number 12934) will be asked to participate in this long term extension study with BAY63-2521.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed 12 weeks of treatment in the double blind trial PATENT 1

Exclusion Criteria:

* Patients who have an ongoing serious adverse event from PATENT 1 that is assessed as related to BAY63-2521 are not allowed to participate in the extension trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2009-03-12 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (91):
- United States (10):
  - Los Angeles, California
  - Sacramento, California
  - Aurora, Colorado
  - Boston, Massachusetts
  - Omaha, Nebraska
  - Cleveland, Ohio
  - Columbus, Ohio
  - Fairfield, Ohio
  - Dallas, Texas
  - El Paso, Texas
- Capital Federal, Argentina
- Australia (5):
  - Darlinghurst, New South Wales
  - Auchenflower, Queensland
  - Herston, Queensland
  - Hobart, Tasmania
  - Prahran, Victoria
- Austria (3):
  - Linz, Upper Austria
  - Innsbruck
  - Vienna
- Belgium (2):
  - Bruxelles - Brussel
  - Leuven
- Brazil (3):
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
  - Rio de Janeiro
- Canada (2):
  - Calgary, Alberta
  - Montreal, Quebec
- China (3):
  - Guangzhou, Guangdong
  - Beijing
  - Shanghai
- Prague, Czechia
- Aarhus N, Denmark
- France (7):
  - Besançon
  - Brest
  - Grenoble
  - Lille
  - Montpellier
  - Pessac
  - Rouen
- Germany (9):
  - Heidelberg, Baden-Wurttemberg
  - München, Bavaria
  - Giessen, Hesse
  - Hanover, Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Cologne, North Rhine-Westphalia
  - Homburg, Saarland
  - Dresden, Saxony
  - Leipzig, Saxony
- Chaïdári, Greece
- Italy (4):
  - Trieste, Friuli Venezia Giulia
  - Rome, Lazio
  - Milan, Lombardy
  - Pavia, Lombardy
- Japan (13):
  - Nagoya, Aichi-ken
  - Kobe, Hyōgo
  - Toride, Ibaraki
  - Tsukuba, Ibaraki
  - Kanazawa, Ishikawa-ken
  - Sendai, Miyagi
  - Tomigusuku, Okinawa
  - Bunkyo-ku, Tokyo
  - Mitaka, Tokyo
  - Ōta-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Hiroshima
  - Okayama
- Mexico (6):
  - Antiguo Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, Jalisco
  - Pulmocritic, Guadalajara, Jalisco
  - Monterrey, Nuevo León
  - Culiacán, Sinaloa
  - Mexico City
  - Querétaro
- Otwock, Poland
- Portugal (3):
  - Coimbra
  - Lisbon
  - Centro Hospitalar de Lisboa Norte - Hospital Santa Maria, Lisbon
- Russia (2):
  - Moscow
  - Saint Petersburg
- Singapore, Singapore
- Seoul, South Korea
- Umeå, Sweden
- Zurich, Switzerland
- Taiwan (2):
  - Kaohsiung City
  - Taipei
- Thailand (2):
  - Bangkok
  - Chiang Mai
- Turkey (Türkiye) (3):
  - Ankara
  - Istanbul
  - Izmir
- United Kingdom (3):
  - Cambridge, Cambridgeshire
  - Clydebank, West Dunbartonshire
  - London

REFERENCES:
- [Background] Benza RL, Boucly A, Farber HW, Frost AE, Ghofrani HA, Hoeper MM, Lambelet M, Rahner C, Bansilal S, Nikkho S, Meier C, Sitbon O. Change in REVEAL Lite 2 risk score predicts outcomes in patients with pulmonary arterial hypertension in the PATENT study. J Heart Lung Transplant. 2022 Mar;41(3):411-420. doi: 10.1016/j.healun.2021.10.013. Epub 2021 Oct 28. PMID 34848133
- [Background] Benza RL, Farber HW, Frost AE, Ghofrani HA, Corris PA, Lambelet M, Nikkho S, Meier C, Hoeper MM. Application of the REVEAL risk score calculator 2.0 in the CHEST study. Respir Med. 2022 Apr-May;195:106783. doi: 10.1016/j.rmed.2022.106783. Epub 2022 Mar 1. PMID 35256218
- [Result] Ghofrani HA, Grimminger F, Grunig E, Huang Y, Jansa P, Jing ZC, Kilpatrick D, Langleben D, Rosenkranz S, Menezes F, Fritsch A, Nikkho S, Humbert M. Predictors of long-term outcomes in patients treated with riociguat for pulmonary arterial hypertension: data from the PATENT-2 open-label, randomised, long-term extension trial. Lancet Respir Med. 2016 May;4(5):361-71. doi: 10.1016/S2213-2600(16)30019-4. Epub 2016 Apr 8. PMID 27067479
- [Result] Ghofrani HA, Humbert M, Langleben D, Schermuly R, Stasch JP, Wilkins MR, Klinger JR. Riociguat: Mode of Action and Clinical Development in Pulmonary Hypertension. Chest. 2017 Feb;151(2):468-480. doi: 10.1016/j.chest.2016.05.024. Epub 2016 Jun 2. PMID 27263466
- [Derived] Benza RL, Ghofrani HA, Grunig E, Hoeper MM, Jansa P, Jing ZC, Kim NH, Langleben D, Simonneau G, Wang C, Busse D, Meier C, Ghio S. Effect of riociguat on right ventricular function in patients with pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension. J Heart Lung Transplant. 2021 Oct;40(10):1172-1180. doi: 10.1016/j.healun.2021.06.020. Epub 2021 Jul 10. PMID 34353714
- [Derived] Humbert M, Coghlan JG, Ghofrani HA, Grimminger F, He JG, Riemekasten G, Vizza CD, Boeckenhoff A, Meier C, de Oliveira Pena J, Denton CP. Riociguat for the treatment of pulmonary arterial hypertension associated with connective tissue disease: results from PATENT-1 and PATENT-2. Ann Rheum Dis. 2017 Feb;76(2):422-426. doi: 10.1136/annrheumdis-2015-209087. Epub 2016 Jul 25. PMID 27457511
- [Derived] Saleh S, Becker C, Frey R, Muck W. Population pharmacokinetics and the pharmacokinetic/pharmacodynamic relationship of riociguat in patients with pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension. Pulm Circ. 2016 Mar;6(Suppl 1):S86-96. doi: 10.1086/685404. PMID 27162632
- [Derived] Rosenkranz S, Ghofrani HA, Beghetti M, Ivy D, Frey R, Fritsch A, Weimann G, Saleh S, Apitz C. Riociguat for pulmonary arterial hypertension associated with congenital heart disease. Heart. 2015 Nov;101(22):1792-9. doi: 10.1136/heartjnl-2015-307832. Epub 2015 Jul 1. PMID 26135803
- [Derived] Rubin LJ, Galie N, Grimminger F, Grunig E, Humbert M, Jing ZC, Keogh A, Langleben D, Fritsch A, Menezes F, Davie N, Ghofrani HA. Riociguat for the treatment of pulmonary arterial hypertension: a long-term extension study (PATENT-2). Eur Respir J. 2015 May;45(5):1303-13. doi: 10.1183/09031936.00090614. Epub 2015 Jan 22. PMID 25614164
- [Derived] Ghofrani HA, Galie N, Grimminger F, Grunig E, Humbert M, Jing ZC, Keogh AM, Langleben D, Kilama MO, Fritsch A, Neuser D, Rubin LJ; PATENT-1 Study Group. Riociguat for the treatment of pulmonary arterial hypertension. N Engl J Med. 2013 Jul 25;369(4):330-40. doi: 10.1056/NEJMoa1209655. PMID 23883378
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 97 centers in 27 countries between 12-MAR-2009 (first participant first visit) and 19-AUG-2019 (last participant last visit);
Pre-assignment Details: Of the 405 participants who completed PATENT-1(NCT00810693) study, 396 participants entered PATENT-2 study. 231 participants were from the former riociguat 1.0-2.5mg group, 109 were from the former placebo group and 56 were from the former riociguat 1.0-1.5mg group.
Groups:
- Riociguat-Former Riociguat 1.0-2.5 mg: Participants from the former riociguat (BAY 63-2521) 1.0 - 2.5 mg treatment group in PATENT-1 on the same dose as they received on the last day of PATENT-1.
- Riociguat-Former Placebo: Participants were from the former placebo group of PATENT-1. The starting dose in PATENT-2 was 1.0 mg riociguat three times one day.
- Riociguat-Former Riociguat 1.0-1.5 mg: Participants from the former riociguat (BAY 63-2521) 1.0 - 1.5 mg treatment group in PATENT-1 on the same dose as they received on the last day of PATENT-1.
Period: Overall Study
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Started | 231 | 109 | 56
Completed | 140 (Completed treatment) | 66 (Completed treatment) | 38 (Completed treatment)
Not Completed | 91 | 43 | 18
Not completed — Other | 2 | 0 | 0
Not completed — Missing | 1 | 0 | 0
Not completed — Death | 40 | 23 | 6
Not completed — Withdrawal by Subject | 12 | 5 | 2
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 3
Not completed — Adverse Event | 28 | 10 | 6
Not completed — Lack of Efficacy | 2 | 2 | 1
Not completed — Non-compliance with study drug | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: All 396 participants who received 1 of 3 blinded treatments for 12 weeks in the double blind PATENT-1 study entered long term extension PATENT-2 study. Baseline of PATENT-2 was Week 0 of PATENT-1. All 396 participants were included in the long term safety set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg | Total
Number analyzed (Participants) | 231 | 109 | 56 | 396
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 174 | 87 | 45 | 306
  >=65 years | 57 | 22 | 11 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (16.4) | 48.8 (15.9) | 48.2 (16.3) | 49.7 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186 | 87 | 44 | 317
  Male | 45 | 22 | 12 | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 148 | 66 | 28 | 242
  Black or African American | 2 | 1 | 1 | 4
  Asian | 74 | 33 | 20 | 127
  Hispanic or Latino | 7 | 8 | 7 | 22
  Multiple | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Description: Analyses of drug-related TEAEs were based on the assessment of causal relationship to study medication.
Time Frame: From administration of first dose of study medication in PATENT-2 up to 2 days after end of treatment with study medication, up to 10 years and 5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 231 | 109 | 56
Participants
  Any TEAE | 229 | 108 | 56
  Any drug-related TEAE | 138 | 74 | 30
  Any serious TEAE | 161 | 76 | 39
  Any drug-related serious TEAE | 25 | 16 | 3
  Any TEAE leading to death | 42 | 25 | 6

2. Primary Outcome: Number of Participant With Death
Description: Analyses of deaths were based on the assessment of causal relationship to study medication. The safety follow-up visit was to be performed 30 days after the last dose of riociguat.
Time Frame: From baseline to end of safety follow-up visit, up to 10 years and 6 months (1 month more than End of study visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 231 | 109 | 56
Participants | 48 | 30 | 7

3. Secondary Outcome: Percentage of Participants With Treatment-emergent High Laboratory Abnormalities in Hematology and Coagulation
Description: Percentage of participants only with a treatment-emergent shift in hematology and coagulation parameters from normal or low at baseline to a high value at a timepoint after the start of treatment. The percentage was calculated by comparing the number of participants with a normal or low value at baseline who had at least one high value after the start of treatment with the number of participants with a normal or low value at baseline who also had at least one valid value after start of treatment.
  A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit, and for each parameter.
Measure: Number; unit: Percentage of participants
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 209 | 93 | 49
Percentage of participants
  aPTT (Sec): number analyzed (Participants) | 94 | 40 | 24
  aPTT (Sec) | 68.1 | 80.0 | 79.2
  Basophils (Giga/L): number analyzed (Participants) | 209 | 91 | 49
  Basophils (Giga/L) | 1.0 | 1.1 | 2.0
  Basophils/Leukocytes (%): number analyzed (Participants) | 207 | 91 | 49
  Basophils/Leukocytes (%) | 16.4 | 12.1 | 10.4
  Eosinophils (Giga/L): number analyzed (Participants) | 208 | 91 | 49
  Eosinophils (Giga/L) | 1.9 | 2.2 | 2.0
  Eosinophils/Leukocytes (%): number analyzed (Participants) | 206 | 89 | 48
  Eosinophils/Leukocytes (%) | 8.7 | 3.4 | 10.4
  Erythrocytes (T/L): number analyzed (Participants) | 190 | 87 | 40
  Erythrocytes (T/L) | 13.7 | 21.8 | 35.0
  Hematocrit (%): number analyzed (Participants) | 163 | 69 | 35
  Hematocrit (%) | 35.6 | 37.7 | 48.6
  Hemoglobin (g/dL): number analyzed (Participants) | 202 | 85 | 45
  Hemoglobin (g/dL) | 8.9 | 16.5 | 24.4
  Leukocytes (Giga/L): number analyzed (Participants) | 202 | 88 | 45
  Leukocytes (Giga/L) | 10.9 | 13.6 | 22.2
  Lymphocytes (Giga/L): number analyzed (Participants) | 209 | 89 | 49
  Lymphocytes (Giga/L) | 1.4 | 3.4 | 0.0
  Lymphocytes/Leukocytes (%): number analyzed (Participants) | 201 | 87 | 46
  Lymphocytes/Leukocytes (%) | 11.4 | 19.5 | 6.5
  Monocytes (Giga/L): number analyzed (Participants) | 205 | 91 | 48
  Monocytes (Giga/L) | 6.3 | 3.3 | 0.0
  Monocytes/Leukocytes (%): number analyzed (Participants) | 205 | 89 | 45
  Monocytes/Leukocytes (%) | 20.0 | 18.0 | 22.2
  Neutrophils (Giga/L): number analyzed (Participants) | 197 | 85 | 46
  Neutrophils (Giga/L) | 14.2 | 18.8 | 28.3
  Neutrophils/Leukocytes (%): number analyzed (Participants) | 186 | 81 | 44
  Neutrophils/Leukocytes (%) | 42.5 | 38.3 | 52.3
  Platelets (Giga/L): number analyzed (Participants) | 201 | 93 | 45
  Platelets (Giga/L) | 14.9 | 9.7 | 15.6
  Prothrombin INR: number analyzed (Participants) | 112 | 50 | 29
  Prothrombin INR | 56.3 | 74.0 | 58.6

4. Secondary Outcome: Percentage of Participants With Treatment-emergent Low Laboratory Abnormalities in Hematology and Coagulation
Description: Percentage of participants only with a treatment-emergent shift in hematology and coagulation parameters from normal or high at baseline to a low value at a timepoint after the start of treatment. The percentage was calculated by comparing the number of participants with a normal or high value at baseline who had at least one low value after the start of treatment with the number of participants with a normal or high value at baseline who also had at least one valid value after start of treatment.
  A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit, and for each parameter.
Measure: Number; unit: Percentage of participants
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 211 | 96 | 49
Percentage of participants
  aPTT (Sec): number analyzed (Participants) | 211 | 96 | 47
  aPTT (Sec) | 12.8 | 13.5 | 8.5
  Erythrocytes (T/L): number analyzed (Participants) | 174 | 79 | 44
  Erythrocytes (T/L) | 31.0 | 22.8 | 25.0
  Hematocrit (%): number analyzed (Participants) | 195 | 90 | 45
  Hematocrit (%) | 22.1 | 23.3 | 26.7
  Hemoglobin (g/dL): number analyzed (Participants) | 170 | 79 | 39
  Hemoglobin (g/dL) | 48.2 | 38.0 | 46.2
  Leukocytes (Giga/L): number analyzed (Participants) | 191 | 89 | 43
  Leukocytes (Giga/L) | 25.7 | 23.6 | 25.6
  Lymphocytes (Giga/L): number analyzed (Participants) | 184 | 82 | 46
  Lymphocytes (Giga/L) | 29.3 | 29.3 | 32.6
  Lymphocytes/Leukocytes (%): number analyzed (Participants) | 169 | 74 | 42
  Lymphocytes/Leukocytes (%) | 50.3 | 44.6 | 64.3
  Monocytes (Giga/L): number analyzed (Participants) | 209 | 91 | 49
  Monocytes (Giga/L) | 0.5 | 1.1 | 2.0
  Monocytes/Leukocytes (%): number analyzed (Participants) | 209 | 91 | 49
  Monocytes/Leukocytes (%) | 2.4 | 3.3 | 14.3
  Neutrophils (Giga/L): number analyzed (Participants) | 203 | 90 | 47
  Neutrophils (Giga/L) | 9.4 | 4.4 | 8.5
  Neutrophils/Leukocytes (%): number analyzed (Participants) | 204 | 88 | 46
  Neutrophils/Leukocytes (%) | 6.9 | 4.5 | 6.5
  Platelets (Giga/L): number analyzed (Participants) | 168 | 78 | 41
  Platelets (Giga/L) | 23.8 | 29.5 | 26.8
  Prothrombin INR: number analyzed (Participants) | 205 | 96 | 46
  Prothrombin INR | 0.0 | 0.0 | 0.0

5. Secondary Outcome: Percentage of Participants With Treatment-emergent High Laboratory Abnormalities in Clinical Chemistry
Description: Percentage of participants per treatment group only with a treatment-emergent shift in clinical chemistry parameters from normal or low at baseline to a high value at a timepoint after the start of treatment. The percentage was calculated by comparing the number of participants with a normal or low value at baseline who had at least one high value after the start of treatment with the number of participants with a normal or low value at baseline who also had at least one valid value after start of treatment.
  A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit, and for each parameter.
Measure: Number; unit: Percentage of participants
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 222 | 103 | 52
Percentage of participants
  Alanine Aminotransferase (U/L): number analyzed (Participants) | 202 | 92 | 46
  Alanine Aminotransferase (U/L) | 13.4 | 12.0 | 8.7
  Albumin (g/dL): number analyzed (Participants) | 222 | 102 | 52
  Albumin (g/dL) | 0.5 | 1.0 | 0.0
  Alkaline Phosphatase (U/L): number analyzed (Participants) | 197 | 94 | 45
  Alkaline Phosphatase (U/L) | 15.7 | 23.4 | 15.6
  Aspartate Aminotransferase (U/L): number analyzed (Participants) | 199 | 96 | 47
  Aspartate Aminotransferase (U/L) | 11.6 | 11.5 | 10.6
  Bilirubin (mg/dL): number analyzed (Participants) | 193 | 93 | 45
  Bilirubin (mg/dL) | 14.5 | 11.8 | 28.9
  Calcium(mg/dL): number analyzed (Participants) | 40 | 15 | 6
  Calcium(mg/dL) | 2.5 | 0.0 | 0.0
  Creatine Kinase (U/L): number analyzed (Participants) | 214 | 97 | 47
  Creatine Kinase (U/L) | 23.8 | 24.7 | 19.1
  Creatinine (mg/dL): number analyzed (Participants) | 160 | 78 | 33
  Creatinine (mg/dL) | 29.4 | 39.7 | 45.5
  Gamma Glutamyl Transferase(U/L): number analyzed (Participants) | 176 | 76 | 40
  Gamma Glutamyl Transferase(U/L) | 18.2 | 17.1 | 25.0
  Glutamate Dehydrogenase (U/L): number analyzed (Participants) | 160 | 69 | 37
  Glutamate Dehydrogenase (U/L) | 40.0 | 37.7 | 56.8
  Phosphate (mg/dL): number analyzed (Participants) | 38 | 14 | 6
  Phosphate (mg/dL) | 2.6 | 0.0 | 0.0
  Potassium (mmol/L): number analyzed (Participants) | 218 | 102 | 50
  Potassium (mmol/L) | 4.6 | 4.9 | 8.0
  Protein (g/dL): number analyzed (Participants) | 216 | 102 | 52
  Protein (g/dL) | 2.3 | 4.9 | 3.8
  Pseudocholinesterase (U/mL): number analyzed (Participants) | 220 | 102 | 52
  Pseudocholinesterase (U/mL) | 0.5 | 0.0 | 0.0
  Sodium (mmol/L) | 0.5 | 1.9 | 3.8
  Triacylglycerol Lipase (U/L): number analyzed (Participants) | 199 | 88 | 49
  Triacylglycerol Lipase (U/L) | 22.6 | 19.3 | 12.2
  Urate (mg/dL): number analyzed (Participants) | 173 | 75 | 41
  Urate (mg/dL) | 24.3 | 25.3 | 29.3
  Urea (mg/dL): number analyzed (Participants) | 199 | 90 | 46
  Urea (mg/dL) | 20.1 | 18.9 | 30.4
  eGFR - MDRD Method (mL/min/1.73 m*2) | 0.0 | 0.0 | 0.0
  Creatinine Clearance (mL/min): number analyzed (Participants) | 198 | 91 | 45
  Creatinine Clearance (mL/min) | 12.1 | 15.4 | 13.3

6. Secondary Outcome: Percentage of Participants With Treatment-emergent Low Laboratory Abnormalities in Clinical Chemistry
Description: Percentage of participants per treatment group only with a treatment-emergent shift in clinical chemistry parameters from normal or high at baseline to a low value at a timepoint after the start of treatment. The percentage was calculated by comparing the number of participants with a normal or high value at baseline who had at least one low value after the start of treatment with the number of participants with a normal or high value at baseline who also had at least one valid value after start of treatment.
  A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit, and for each parameter.
Measure: Number; unit: Percentage of participants
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 223 | 103 | 52
Percentage of participants
  Alanine Aminotransferase (U/L): number analyzed (Participants) | 1 | 1 | 1
  Alanine Aminotransferase (U/L) | 0.0 | 0.0 | 0.0
  Albumin (g/dL): number analyzed (Participants) | 221 | 101 | 51
  Albumin (g/dL) | 4.1 | 4.0 | 0.0
  Alkaline Phosphatase (U/L): number analyzed (Participants) | 215 | 101 | 51
  Alkaline Phosphatase (U/L) | 3.3 | 4.0 | 0.0
  Bilirubin (mg/dL) | 0.0 | 1.0 | 0.0
  Calcium (mg/dL): number analyzed (Participants) | 40 | 10 | 5
  Calcium (mg/dL) | 25.0 | 10.0 | 20.0
  Creatine Kinase (U/L): number analyzed (Participants) | 207 | 99 | 49
  Creatine Kinase (U/L) | 8.7 | 5.1 | 12.2
  Creatinine (mg/dL): number analyzed (Participants) | 221 | 102 | 52
  Creatinine (mg/dL) | 4.5 | 6.9 | 5.8
  Gamma Glutamyl Transferase (U/L): number analyzed (Participants) | 222 | 103 | 52
  Gamma Glutamyl Transferase (U/L) | 0.0 | 0.0 | 0.0
  Phosphate (mg/dL): number analyzed (Participants) | 38 | 13 | 6
  Phosphate (mg/dL) | 5.3 | 15.4 | 33.3
  Potassium (mmol/L): number analyzed (Participants) | 213 | 95 | 47
  Potassium (mmol/L) | 24.9 | 32.6 | 29.8
  Protein (g/dL): number analyzed (Participants) | 211 | 97 | 47
  Protein (g/dL) | 9.0 | 10.3 | 8.5
  Pseudocholinesterase (U/mL): number analyzed (Participants) | 209 | 99 | 50
  Pseudocholinesterase (U/mL) | 11.0 | 11.1 | 8.0
  Sodium (mmol/L): number analyzed (Participants) | 213 | 100 | 51
  Sodium (mmol/L) | 8.5 | 13.0 | 11.8
  Triacylglycerol Lipase (U/L): number analyzed (Participants) | 222 | 103 | 52
  Triacylglycerol Lipase (U/L) | 0.0 | 0.0 | 0.0
  Urate (mg/dL): number analyzed (Participants) | 222 | 101 | 52
  Urate (mg/dL) | 3.6 | 5.0 | 3.8
  Urea (mg/dL): number analyzed (Participants) | 222 | 103 | 52
  Urea (mg/dL) | 0.9 | 1.0 | 0.0
  eGFR - MDRD Method(mL/min/1.73 m*2): number analyzed (Participants) | 179 | 86 | 43
  eGFR - MDRD Method(mL/min/1.73 m*2) | 19.0 | 17.4 | 23.3
  Creatinine Clearance (mL/min): number analyzed (Participants) | 127 | 66 | 31
  Creatinine Clearance (mL/min) | 45.7 | 30.3 | 48.4

7. Other Pre Specified Outcome: Change of Systolic Blood Pressure (SBP)
Description: SBP was measured after the participant had been at rest for 10 minutes in a supine position. Low SBP was defined as SBP <95 mmHg, normal SBP as SBP 95-140mmHg, and high SBP as SBP >140 mmHg.
  A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: millimetre(s) of mercury (mmHg)
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 231 | 109 | 56
millimetre(s) of mercury (mmHg)
  Baseline (Week 0) | 114.36 (14.78) | 113.75 (12.76) | 110.88 (12.49)
  Change from baseline to Termination visit: number analyzed (Participants) | 169 | 80 | 41
  Change from baseline to Termination visit | -0.88 (15.82) | -1.30 (15.62) | -0.99 (16.12)

8. Other Pre Specified Outcome: Change of Diastolic Blood Pressure (DBP)
Description: DBP was measured after the participants had been at rest for 10 minutes in a supine position.
  A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 231 | 109 | 56
mmHg
  Baseline (Week 0) | 72.03 (10.53) | 71.84 (9.06) | 69.61 (9.89)
  Change from baseline to Termination visit: number analyzed (Participants) | 169 | 80 | 41
  Change from baseline to Termination visit | -3.33 (12.90) | -4.00 (11.72) | -2.13 (9.65)

9. Other Pre Specified Outcome: Change of Heart Rate
Description: Heart rate was measured after the participant had been at rest for 10 minutes in a supine position.
  A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: beats/minute (BPM)
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 231 | 109 | 56
beats/minute (BPM)
  Baseline (Week 0) | 76.47 (11.04) | 77.30 (12.53) | 76.04 (10.83)
  Change from baseline to Termination visit: number analyzed (Participants) | 169 | 80 | 41
  Change from baseline to Termination visit | 0.75 (13.92) | 0.18 (14.07) | -1.10 (14.74)

10. Other Pre Specified Outcome: Change of Weight
Description: Weight was evaluated for safety. A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 231 | 109 | 56
kilogram (kg)
  Baseline (Week 0) | 68.24 (18.25) | 69.03 (16.94) | 69.57 (14.69)
  Change from baseline to Termination visit: number analyzed (Participants) | 169 | 81 | 41
  Change from baseline to Termination visit | -1.67 (6.45) | 0.04 (6.04) | -1.79 (8.08)

11. Other Pre Specified Outcome: Change of Oxygen Saturation (SaO2)
Description: SaO2 is one parameters of blood gas. The sample was obtained with the participant resting in a sitting or supine position for at least 10 minutes.
  A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 227 | 109 | 56
Percentage
  Baseline (Week 0) | 95.10 (2.61) | 94.32 (3.18) | 94.00 (2.95)
  Change from baseline to Termination visit: number analyzed (Participants) | 15 | 9 | 2
  Change from baseline to Termination visit | -1.14 (3.48) | -0.56 (4.45) | -4.30 (5.23)

12. Other Pre Specified Outcome: Change of Arterial Partial Oxygen Pressure (PaO2)
Description: PaO2 is one parameter of blood gas. The sample was obtained with the participant resting in a sitting or supine position for at least 10 minutes.
  A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 227 | 109 | 56
mmHg
  Baseline (Week 0) | 76.99 (17.60) | 74.54 (17.84) | 72.12 (13.63)
  Change from baseline to Termination visit: number analyzed (Participants) | 15 | 9 | 2
  Change from baseline to Termination visit | -4.77 (17.42) | 7.14 (58.00) | -8.05 (2.76)

13. Other Pre Specified Outcome: Change of Arterial Partial Pressure of Carbon Dioxide (PaCO2)
Description: PaCO2 is one parameter of blood gas. The sample was obtained with the participant resting in a sitting or supine position for at least 10 minutes.
  A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to termination visit, up to 10 years
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 227 | 109 | 56
mmHg
  Baseline (Week 0) | 32.94 (4.62) | 32.46 (4.63) | 33.40 (4.41)
  Change from baseline to Termination visit: number analyzed (Participants) | 15 | 9 | 2
  Change from baseline to Termination visit | -1.87 (3.72) | -0.68 (5.70) | 2.00 (4.24)

14. Other Pre Specified Outcome: Change of RR Duration From Electrocardiogram (ECG)
Description: Heart rate from ECG is derived from the RR duration, unless arrhythmias such as atrial fibrillation or ventricular extra beats require additional calculations. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position.
  Analyses up to Month 48. After this timepoint, data was available for considerably fewer participants in the analysis set.
Time Frame: From baseline to Month 48
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 218 | 103 | 53
millisecond (msec)
  Baseline (Week 0) | 817.69 (125.61) | 828.96 (146.32) | 822.33 (130.27)
  Change from baseline to Month 48: number analyzed (Participants) | 15 | 7 | 6
  Change from baseline to Month 48 | 59.07 (109.89) | 75.69 (181.94) | 89.61 (113.25)

15. Other Pre Specified Outcome: Change of PR Duration From ECG
Description: PR duration was evaluated as part of ECG. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position.
  Analyses up to Month 48. After this timepoint, data was available for considerably fewer participants in the analysis set.
Time Frame: From baseline to Month 48
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 211 | 102 | 53
msec
  Baseline (Week 0) | 171.07 (27.76) | 173.97 (32.90) | 171.74 (25.77)
  Change from baseline to Month 48: number analyzed (Participants) | 15 | 6 | 6
  Change from baseline to Month 48 | 7.51 (16.29) | 16.50 (19.41) | -3.22 (17.18)

16. Other Pre Specified Outcome: Change of QRS Duration From ECG
Description: QRS duration was evaluated as part of ECG. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position.
  Analyses up to Month 48. After this timepoint, data was available for considerably fewer participants in the analysis set.
Time Frame: From baseline to Month 48
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 213 | 103 | 53
msec
  Baseline (Week 0) | 99.59 (17.38) | 100.09 (16.15) | 103.22 (19.82)
  Change from baseline to Month 48: number analyzed (Participants) | 15 | 7 | 6
  Change from baseline to Month 48 | 5.07 (8.56) | 11.14 (18.69) | -0.44 (7.52)

17. Other Pre Specified Outcome: Change of QT Duration in ECG
Description: QT duration was evaluated as part of ECG. ECGs were recorded after the participant had been at rest for 15 minutes in a supine position.
  Analyses up to Month 48. After this timepoint, data was available for considerably fewer participants in the analysis set.
Time Frame: From baseline to Month 48
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 177 | 76 | 40
msec
  Baseline (Week 0) | 401.56 (31.35) | 406.67 (35.44) | 405.10 (30.52)
  Change from baseline to Month 48: number analyzed (Participants) | 9 | 3 | 4
  Change from baseline to Month 48 | 10.93 (27.58) | 16.89 (16.78) | 27.34 (28.61)

18. Other Pre Specified Outcome: Change in Six-minute Walking Distance (6MWD) Test
Description: 6MWD is exercise testing and is one of efficacy evaluation
Time Frame: From baseline to End of study visit, up to 10 years and 5 months.
Measure: Median (Full Range); unit: meters
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 231 | 109 | 56
meters
  Baseline (Week 0) | 375.0 (160) [160 to 468] | 395.0 (174) [174 to 450] | 376.0 (158) [158 to 448]
  Change from baseline to End of study visit | 19.0 (-448) [-448 to 309] | 9.0 (-446) [-446 to 275] | 1.5 (-448) [-448 to 492]

19. Other Pre Specified Outcome: Change in Pulmonary Vascular Resistance (PVR)
Description: Pulmonary vascular resistance (PVR) was measured only if right-heart catheterization was performed as part of a regular diagnostic work-up.
  A termination visit was only to be performed in the case of premature termination of study medication or if the sponsor announced the official end of the study.
Time Frame: From baseline to Termination visit, up to 10 years 5 months
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: dyn*s*cm^-5
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 228 | 103 | 56
dyn*s*cm^-5
  Baseline (Week 0) | 802.40 (452.97) | 835.45 (476.52) | 855.70 (552.92)
  Change from baseline to Termination visit: number analyzed (Participants) | 2 | 0 | 0
  Change from baseline to Termination visit | 34.25 (104.83) |  |

20. Other Pre Specified Outcome: Change in N-terminal Prohormone of Brain Natriuretic Peptide (NT-proBNP)
Description: NT-proBNP levels in the blood are used for diagnosis of acute congestive heart failure (CHF) and may be useful to establish prognosis in heart failure
Time Frame: From baseline to End of study visit, up to 10 year and 5 months
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: picograms/millilitre (pg/mL)
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 210 | 97 | 47
picograms/millilitre (pg/mL)
  Baseline (Week 0) | 996.30 (1627.48) | 1135.68 (1533.20) | 1220.11 (1457.90)
  Change from baseline to End of study visit | 82.52 (2253.30) | 202.42 (3466.94) | 115.77 (1918.81)

21. Other Pre Specified Outcome: Change in World Health Organization (WHO) Functional Class
Description: WHO classification: I: Participants with PH. Ordinary physical activity does not cause undue dyspnea or fatigue, chest pain, or near syncope. II: Participants with PH are comfortable at rest. Ordinary physical activity causes undue dyspnea or fatigue, chest pain, or near syncope. III: Participants with PH are comfortable at rest. Less than ordinary activity causes undue dyspnea or fatigue, chest pain, or near syncope. IV: Participants with PH with inability to carry out any physical activity. They manifest signs of right-heart failure. Dyspnea and/or fatigue may even be present at rest. For class change from baseline, minus indicates a participant's functional class decreased compared with baseline (e.g. "-1" indicates a participant changed from class IV to class III, or from class II to class I), plus indicates a participant's functional class increased compared with baseline (e.g. "+1" indicates a participant changed from class I to class II, or from class III to class IV).
Time Frame: From baseline to End of study visit, up to 10 years and 5 months.
Population: Participants in SAF with evaluable data for each visit
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 231 | 109 | 56
Participants
  Baseline (Week 0)-class I | 5 | 3 | 4
  Baseline (Week 0)-class II | 98 | 54 | 17
  Baseline (Week 0)-class III | 128 | 49 | 35
  Baseline (Week 0)-class IV | 0 | 2 | 0
  Baseline (Week 0)-Missing | 0 | 1 | 0
  Change from baseline to EOS visit- -2: number analyzed (Participants) | 231 | 108 | 56
  Change from baseline to EOS visit- -2 | 5 | 0 | 1
  Change from baseline to EOS visit- -1: number analyzed (Participants) | 231 | 108 | 56
  Change from baseline to EOS visit- -1 | 50 | 16 | 13
  Change from baseline to EOS visit- 0: number analyzed (Participants) | 231 | 108 | 56
  Change from baseline to EOS visit- 0 | 101 | 52 | 28
  Change from baseline to EOS visit- +1: number analyzed (Participants) | 231 | 108 | 56
  Change from baseline to EOS visit- +1 | 23 | 15 | 6
  Change from baseline to EOS visit- +2: number analyzed (Participants) | 231 | 108 | 56
  Change from baseline to EOS visit- +2 | 33 | 17 | 5
  Change from baseline to EOS visit- +3: number analyzed (Participants) | 231 | 108 | 56
  Change from baseline to EOS visit- +3 | 19 | 8 | 3

22. Other Pre Specified Outcome: Number of Participants With Clinical Worsening
Description: Time to clinical worsening was a parameter that combined death and events reflective of persistent clinical worsening of the participant's underlying diagnosis of pulmonary hypertension (PH)
Time Frame: From baseline to End of study visit, up to 10 years and 5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 231 | 109 | 56
Participants
  Any clinical worsening | 87 | 41 | 18
  Heart/lung transplantation | 3 | 0 | 2
  Atrial septostomy | 1 | 1 | 0
  Hospitalization due to pulmonary hypertension | 29 | 12 | 8
  Start of new pulmonary hypertension treatment | 52 | 20 | 14
  Decrease in 6MWD due to pulmonary hypertension | 7 | 6 | 2
  Persistent worsening of functional class due to PH | 8 | 2 | 1
  Death | 48 | 30 | 7

23. Other Pre Specified Outcome: Incidence of Clinical Worsening Events Per 100 Person Years
Description: as for outcome 22
Time Frame: From baseline to End of study visit, up to 10 years and 5 months.
Measure: Number; unit: Percentage per 100 person-years
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 231 | 109 | 56
Percentage per 100 person-years
  Any clinical worsening event | 22.09 | 22.10 | 19.20
  Heart/Lung Transplantation | 0.34 | 0 | 0.89
  Atrial Septostomy | 0.11 | 0.25 | 0
  Hospitalization due to PH | 4.46 | 3.81 | 5.80
  Start of new PH treatment | 9.73 | 8.13 | 7.59
  Decrease in 6MWD due to PH | 1.03 | 1.78 | 0.89
  Persistent worsening of functional class due to PH | 0.92 | 0.51 | 0.89
  Death | 5.49 | 7.62 | 3.13

24. Other Pre Specified Outcome: Change From Baseline in Borg CR 10 Scale
Description: The Borg CR10 Scale was measured in conjunction with the 6MWD test. The test was explained to the participant before starting the 6MWD test. Participants were asked to rank their exertion at the end of the 6MWD test. Low values indicate low levels of exertion; high values indicate more intense exertion reported by the participant. The score ranges from 0 ("Nothing at all") to 10 ("Extremely strong - Maximal")
Time Frame: From baseline to Week 12
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 231 | 109 | 56
Scores on a scale
  Baseline (Week 0) | 3.87 (2.24) | 3.80 (2.26) | 3.41 (1.77)
  Change from baseline to Week 12: number analyzed (Participants) | 216 | 101 | 54
  Change from baseline to Week 12 | -0.58 (1.84) | -0.54 (1.91) | -0.52 (1.64)

25. Other Pre Specified Outcome: Change in Score of EQ-5D Questionnaire
Description: The EQ-5D is a standardized instrument for use as a measure of health outcome. The EQ-5D is a self report questionnaire. The utility score is calculated based on five questions concerning problems with mobility, self-care, usual activities, pain/discomfort and anxiety/depression. An increase in the utility score represents an improvement in quality of life. The score ranges from -0.594 (worst answer in all five questions) to 1 (best answer in all five questions).
Time Frame: From baseline to End of study visit, up to 10 years and 5 months.
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 230 | 107 | 55
Scores on a scale
  Baseline (Week 0) | 0.6883 (0.2339) | 0.6929 (0.2302) | 0.6338 (0.2744)
  Change from baseline to EOS Visit | -0.2452 (0.5894) | -0.2812 (0.5944) | -0.0925 (0.4376)

26. Other Pre Specified Outcome: Change in Score of Living With Pulmonary Hypertension (LPH) Questionnaire
Description: The LPH questionnaire is designed to measure the effects of PH and PH-specific treatments on an individual's quality of life. The LPH is a self-report questionnaire and was completed by the participant. The LPH total score can range from 0 (best) to 105 (worst).
Time Frame: From baseline to End of study visit, up to 10 years and 5 months.
Population: Participants in SAF with evaluable data for each visit
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat-Former Riociguat 1.0-2.5 mg | Riociguat-Former Placebo | Riociguat-Former Riociguat 1.0-1.5 mg
Number analyzed (Participants) | 225 | 105 | 55
Scores on a scale
  Baseline (Week 0) | 41.77 (22.18) | 41.94 (23.34) | 45.10 (22.08)
  Change from baseline to EOS Visit | 4.99 (34.04) | 12.28 (32.76) | -4.07 (31.40)

ADVERSE EVENTS:
Time Frame: From administration of first dose of study medication in PATENT-2 up to 2 days after end of treatment with study medication, up to 10 years and 5 months.
Groups:
- Former Riociguat 1.0- 2.5 mg: Patients from the PATENT-1 1.0 - 2.5 mg Dose Arm will enter the extension trial (PATENT-2)with the same dose which they have received on the last day of PATENT-1 (Visit 6).
- Former Riociguat 1.0 - 1.5 mg: Patients from the PATENT-1 1.0 - 1.5 mg Dose Arm will enter the extension trial (PATENT-2)with the same dose which they have received on the last day of PATENT-1 (Visit 6).
- Former Placebo: Patients from the PATENT-1 Placebo Arm will enter the extension trial (PATENT-2)with the starting dose 1 mg Riociguat tid.
Arm/Group | Former Riociguat 1.0- 2.5 mg | Former Riociguat 1.0 - 1.5 mg | Former Placebo
All-Cause Mortality (participants affected / at risk) | 48/231 | 7/56 | 30/109
Serious Adverse Events (participants affected / at risk) | 161/231 | 39/56 | 76/109
Other Adverse Events (participants affected / at risk) | 218/231 | 54/56 | 106/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Former Riociguat 1.0- 2.5 mg (N=231) | Former Riociguat 1.0 - 1.5 mg (N=56) | Former Placebo (N=109)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 1 (1) | 6 (7)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 3 (3) | 1 (1) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2)
Atrial flutter (Cardiac disorders) | 5 (5) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 8 (13) | 1 (3) | 7 (8)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (4) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cor pulmonale chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 26 (47) | 7 (9) | 6 (8)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Cardiac dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Heart disease congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (2) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Choroidal neovascularisation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Optic nerve disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (5) | 1 (1) | 1 (2)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastritis haemorrhagic (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 2 (2)
Death (General disorders) | 2 (2) | 0 (0) | 3 (3)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 2 (3)
Sudden death (General disorders) | 2 (2) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 2 (2)
Exercise tolerance decreased (General disorders) | 1 (1) | 0 (0) | 0 (0)
Drug intolerance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular stent stenosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic congestion (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 5 (5) | 2 (3) | 2 (4)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (3) | 0 (0)
Cervicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endometritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 3 (4)
Gastroenteritis (Infections and infestations) | 7 (7) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Infected skin ulcer (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 6 (7) | 7 (9)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 4 (5) | 2 (2) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Appendiceal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ureteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastric infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
Serratia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Systemic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (4)
Brain herniation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Biopsy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Catheterisation cardiac (Investigations) | 18 (24) | 3 (3) | 4 (4)
Chest X-ray abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Endoscopy (Investigations) | 1 (1) | 2 (2) | 0 (0)
Endoscopy upper gastrointestinal tract (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transplant evaluation (Investigations) | 1 (2) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 2 (5) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lymphatic system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Coma hepatic (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 26 (43) | 5 (5) | 15 (23)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Brain stem syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Central nervous system vasculitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 4 (4) | 0 (0) | 2 (2)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 1 (2) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Endometrial dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diaphragm muscle weakness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 2 (2) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 6 (8) | 6 (8)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary veno-occlusive disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal cavity mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 31 (50) | 11 (13) | 14 (28)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fixed eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0)
Homicide (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Atrial septal defect repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel decompression (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Gastric polypectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Lung transplant (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Osteotomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Prophylaxis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Swan ganz catheter placement (Surgical and medical procedures) | 2 (3) | 0 (0) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Dental operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Varicose vein operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (2)
Bladder polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 1 (2) | 0 (0) | 0 (0)
Balloon atrial septostomy (Surgical and medical procedures) | 1 (2) | 1 (1) | 0 (0)
Trapeziectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 5 (5) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Lead dislodgement (Product Issues) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Former Riociguat 1.0- 2.5 mg (N=231) | Former Riociguat 1.0 - 1.5 mg (N=56) | Former Placebo (N=109)
Anaemia (Blood and lymphatic system disorders) | 30 (35) | 6 (6) | 14 (29)
Atrioventricular block first degree (Cardiac disorders) | 3 (3) | 3 (3) | 3 (3)
Cardiac failure (Cardiac disorders) | 6 (6) | 4 (4) | 2 (2)
Palpitations (Cardiac disorders) | 22 (27) | 5 (9) | 14 (14)
Right ventricular failure (Cardiac disorders) | 7 (10) | 3 (3) | 6 (6)
Tachycardia (Cardiac disorders) | 9 (10) | 4 (7) | 4 (6)
Vertigo (Ear and labyrinth disorders) | 6 (6) | 1 (1) | 6 (7)
Abdominal distension (Gastrointestinal disorders) | 14 (20) | 0 (0) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 17 (24) | 4 (4) | 9 (11)
Abdominal pain upper (Gastrointestinal disorders) | 18 (19) | 2 (2) | 7 (8)
Constipation (Gastrointestinal disorders) | 22 (26) | 2 (2) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 50 (81) | 11 (22) | 34 (62)
Dyspepsia (Gastrointestinal disorders) | 34 (68) | 8 (9) | 14 (22)
Gastritis (Gastrointestinal disorders) | 7 (8) | 3 (3) | 10 (12)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 16 (19) | 6 (6) | 13 (16)
Nausea (Gastrointestinal disorders) | 46 (63) | 8 (10) | 26 (41)
Vomiting (Gastrointestinal disorders) | 36 (47) | 9 (19) | 23 (34)
Asthenia (General disorders) | 17 (23) | 3 (4) | 6 (8)
Chest discomfort (General disorders) | 15 (26) | 6 (7) | 6 (6)
Chest pain (General disorders) | 32 (44) | 7 (7) | 16 (25)
Fatigue (General disorders) | 20 (23) | 4 (6) | 12 (20)
Oedema (General disorders) | 9 (11) | 4 (6) | 9 (11)
Oedema peripheral (General disorders) | 64 (108) | 17 (26) | 31 (51)
Pyrexia (General disorders) | 24 (45) | 3 (3) | 7 (8)
Peripheral swelling (General disorders) | 7 (7) | 5 (7) | 4 (5)
Bronchitis (Infections and infestations) | 24 (35) | 11 (13) | 14 (19)
Conjunctivitis (Infections and infestations) | 8 (10) | 3 (5) | 4 (4)
Gastroenteritis (Infections and infestations) | 14 (15) | 6 (6) | 6 (7)
Gastrointestinal infection (Infections and infestations) | 9 (11) | 3 (5) | 3 (3)
Influenza (Infections and infestations) | 14 (21) | 7 (7) | 4 (5)
Lower respiratory tract infection (Infections and infestations) | 8 (11) | 3 (5) | 6 (17)
Nasopharyngitis (Infections and infestations) | 76 (160) | 21 (44) | 31 (81)
Oral candidiasis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 9 (13) | 4 (8) | 4 (4)
Pneumonia (Infections and infestations) | 9 (9) | 7 (7) | 8 (10)
Sinusitis (Infections and infestations) | 13 (25) | 1 (1) | 9 (11)
Upper respiratory tract infection (Infections and infestations) | 39 (64) | 10 (20) | 24 (49)
Urinary tract infection (Infections and infestations) | 12 (21) | 9 (12) | 12 (17)
Lung infection (Infections and infestations) | 4 (5) | 3 (4) | 4 (4)
Respiratory tract infection (Infections and infestations) | 24 (53) | 5 (10) | 13 (19)
Fall (Injury, poisoning and procedural complications) | 12 (13) | 1 (1) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 17 (24) | 1 (1) | 3 (4)
Blood potassium decreased (Investigations) | 8 (10) | 3 (3) | 4 (6)
International normalised ratio increased (Investigations) | 9 (11) | 4 (5) | 4 (4)
Weight decreased (Investigations) | 8 (9) | 0 (0) | 6 (7)
Weight increased (Investigations) | 6 (8) | 5 (7) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 26 (34) | 9 (14) | 12 (16)
Iron deficiency (Metabolism and nutrition disorders) | 11 (13) | 4 (4) | 7 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 (34) | 6 (7) | 10 (15)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 36 (48) | 5 (7) | 11 (17)
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (4) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (4) | 9 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 (16) | 4 (4) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (4) | 7 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 (35) | 7 (7) | 12 (15)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 67 (118) | 15 (22) | 31 (57)
Headache (Nervous system disorders) | 46 (102) | 10 (14) | 34 (61)
Hypoaesthesia (Nervous system disorders) | 9 (9) | 4 (4) | 3 (3)
Presyncope (Nervous system disorders) | 5 (5) | 2 (4) | 8 (9)
Anxiety (Psychiatric disorders) | 10 (10) | 1 (1) | 8 (14)
Depression (Psychiatric disorders) | 13 (13) | 3 (5) | 6 (7)
Insomnia (Psychiatric disorders) | 21 (24) | 5 (5) | 10 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 66 (94) | 13 (20) | 28 (42)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 (54) | 12 (15) | 15 (21)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 30 (42) | 12 (18) | 16 (20)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 20 (46) | 2 (6) | 9 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 3 (4) | 6 (7)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12 (16) | 2 (2) | 8 (10)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 3 (4) | 4 (6)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 15 (20) | 2 (2) | 13 (20)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) | 3 (4)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (5) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (16) | 3 (3) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 13 (18) | 3 (3) | 3 (4)
Haematoma (Vascular disorders) | 7 (8) | 3 (3) | 2 (2)
Hypotension (Vascular disorders) | 32 (39) | 10 (13) | 10 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2012-12-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT00863681/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT00863681/SAP_001.pdf